CLINICAL TRIAL: NCT03896243
Title: Serum Antimullerian Hormone Levels in Patients Who Underwent Uterine Artery Ligation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: uterinarter
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Uterine Artery Ligation; Ovarian Reserve
Keywords: Uterine atony; amh
MeSH Terms: conditions — Uterine Inertia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uterine artery ligation (UAL): We would like toinvite the patients to the hospital at least 6 months after surgery who underwent only uterine artery ligation performed due to uterine atony during C-section.
  They would be evaluated for their ovarian reserve via hormones and antral follicle count (AFC)
  Interventions: Diagnostic Test: Uterine artery ligation (UAL)
- Control Group:: We would like to invite the patients to the hospital at least 6 months after C-section who delivered baby without any complication.
  They would be also evaluated for their ovarian reserve via hormones and antral follicle count (AFC)
  Interventions: Diagnostic Test: Uterine artery ligation (UAL)

INTERVENTIONS:
Diagnostic Test: Uterine artery ligation (UAL) — Uterine artery ligation (UAL) We will invite the patients to the hospital at least 6 months after surgery who underwent only uterine artery ligation performed due to uterine atony during C-section.
  They will evaluated for their ovarian reserve via hormones and antral follicle count (AFC)

SUMMARY:
Investigators would like to see the amh values after uterine artery ligation

DETAILED DESCRIPTION:
Group/cohort:

Uterine artery ligation (UAL) Investigators would like to invite the patients to the hospital at least 6 months after surgery who underwent only uterine artery ligation performed due to uterine atony during C-section.

Participants would be evaluated for their ovarian reserve via hormones and antral follicle count (AFC)

Control Group:

Investigators would like to invite the patients to the hospital at least 6 months after C-section who delivered baby without any complication.

Participants would be also evaluated for their ovarian reserve via hormones and antral follicle count (AFC)

ELIGIBILITY:
Inclusion Criteria:

* age 18- 35 years
* no systemic or endocrine diseases
* patients who had uterine artery ligation due to atony
* healthy postpartum patients as controls

Exclusion Criteria:

* patients with PCOS

  * Pregnancy with IVF or oosit donation
  * Patients with endocrinopathy, diseases which require radiotherapy and chemotherapy etc.
  * Patients with BMI >40

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants are females undergoing delivery of their baby
Study Population: Patients who had uterine artery ligation during C-section. Control group is age-matched postpartum patients.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
1.ovarian reserve in patients with uterine artery ligation | 12 months
  calculation of ovarian reserve with amh (ng/ml) after uterine artery ligation due to uterine atony

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months